CLINICAL TRIAL: NCT05711914
Title: Predicting Response to PD-1 Checkpoint Blockade Using Deep Learning Analysis of Imaging and Clinical Data
Acronym: Onc AI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: MEDEXPRIM (Unknown); GRATICULE (Unknown)
Responsible Party: Sponsor
Other Study IDs: Local2021/JPB-01
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immunotherapy has transformed cancer treatment with the PD-1 class of checkpoint inhibitors - pembrolizumab and nivolumab -- demonstrating durable responses in Stage IV metastatic tumors such as non-small cell lung cancer and melanoma. Despite these numerous successes, PD-1/PD-L1 checkpoint blockade therapies do have a number of shortcomings.

Many approaches to predict response to PD-1/PD-L1 checkpoint therapy have been investigated with limited success. Recent efforts exploring the utility of quantitative imaging biomarkers to predict response to PD-[L]1 immunotherapy have shown promise. The purpose of this retrospective multicenter study is to develop a multi-omic classifier to predict response to PD-1/PD-L1 checkpoint blockade for mutation negative (EGFR, ALK and ROS1) NSCLC

DETAILED DESCRIPTION:
Recent Phase III studies have demonstrated the effectiveness of atezolizumab (PD-L1) in metastatic triple-negative breast cancer [3] and small cell lung cancer, while the standard of care for Stage III non-small cell lung cancer has changed with positive results of the PACIFIC Phase III study, where durvalumab (PD-L1) administered after chemoradiation showed a significant increase in overall survival.

Low response rates, generally in the 15% to 20% range in most diseases when used as a single agent, high therapy cost globally ($150,000 or more per year in the U.S) and serious immune-mediated adverse events, particularly when PD-1/PD-L1 inhibitors are combined with the CTLA-4 inhibitors (ipilimumab). Unpredictable and low patient response rates coupled with high drugs costs and serious toxicities can significantly burden healthcare systems, third-party payers and patients. Clearly, diagnostic tools to stratify patients according to response likelihood are necessary as PD-[L]1 checkpoint inhibitors continue to gain adoption.

The standard-of-care biomarker is an immunohistochemistry (IHC) test that measures levels of the PD-L1 protein expressed in tumor samples. Tumor mutational burden, presence of Tumor-Infiltrating Lymphocytes and inflammatory cytokines are being explored in multiple clinical trials involving PD-(L)1 often in combination with additional immuno-oncology (IO) therapies In such an approach, a non-invasive imaging scan can provide insight and information on the patient's entire tumor burden rather than a sample of a subset of lesions (as provided by biopsy or serum-based assays). When diagnostic images that depict all treatable lesions are further analyzed with computational techniques such as machine-learning and artificial intelligence, resulting in the identification of relevant imaging biomarkers, an accurate overall assessment of patient response to PD-[L]1 therapy may be attainable.

ELIGIBILITY:
Inclusion Criteria:Patients between 18 and 100 years of age -

Exclusion Criteria: Patient under 18 years of age

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with non-small cell lung cancer (NSCLC), having undergone treatment with immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
developing a multi-omic classifier for predicting PD-1 response | during one month
  Once sufficient patient data are accumulated, imaging data (both baseline and follow-up scans) will be annotated (segmented) to delineate lesions, lymph nodes, surrounding organs, etc…

CONTACTS AND LOCATIONS:
Locations (1):
- Jean-Paul BEREGI, Nîmes, France

IPD SHARING:
Plan to Share IPD: No